CLINICAL TRIAL: NCT00002783
Title: A PHASE II TRIAL OF NEOADJUVANT CISPLATIN-FLUOROURACIL CHEMOTHERAPY, SURGERY, AND INTRAPERITONEAL (IP) FLOXURIDINE (FUdR) PLUS LEUCOVORIN IN PATIENTS WITH GASTRIC CANCER
Brief Title: Combination Chemotherapy Before and After Surgery in Treating Patients With Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 96-027; CDR0000064831 (Registry Identifier: PDQ (Physician Data Query)); NCI-H96-0916
Record Dates: First submitted 1999-11-01; First posted 2004-08-24 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Gastric Cancer
Keywords: stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Floxuridine; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: cisplatin
Drug: floxuridine
Drug: fluorouracil
Drug: leucovorin calcium
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them in different ways may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy before and after surgery in treating patients with high-risk stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy and toxicity of neoadjuvant cisplatin/fluorouracil (CDDP/5-FU) followed by surgery followed by adjuvant intraperitoneal floxuridine/leucovorin in patients with high-risk gastric cancer. II. Assess the quality of life and cost-benefit ratio associated with this treatment. III. Evaluate the sensitivity, specificity, and overall staging accuracy of laparoscopy with or without laparoscopic ultrasound in predicting the resectability rate (with and without neoadjuvant CDDP/5-FU), response to chemotherapy, and accuracy when compared to pathologic findings. IV. Correlate the presence of mutated vs. wild-type p53 suppressor oncogenes in endoscopic biopsies and resected tumor specimens with clinical outcome (defined as downstaging, failure pattern, and disease-free and overall survival) in patients treated with and without neoadjuvant CDDP/5-FU.

OUTLINE: The following acronyms are used: CDDP Cisplatin, NSC-119875 CF Leucovorin calcium, NSC-3590 5-FU Fluorouracil, NSC-19893 FUDR Floxuridine, NSC-27640 2-Drug Combination Chemotherapy followed by Surgery followed by Single-Agent Chemotherapy with Drug Modulation. CDDP/5-FU; followed by total or subtotal radical gastrectomy with D2 dissection; followed by FUDR; with CF.

PROJECTED ACCRUAL: A total of 50 patients will be entered over 2-2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Microscopically confirmed adenocarcinoma of the stomach or gastroesophageal junction Reviewed by Department of Pathology of participating institution Stage II-IV (T2, N1-2, M0 or T3-4, any N, M0) by physical exam, CT, and laparoscopy Potentially curable by surgery Suspected sites of metastasis proven M0 prior to entry

PATIENT CHARACTERISTICS: Age: Any age Performance status: Karnofsky 60%-100% Hematopoietic: WBC at least 4,000 Platelets at least 150,000 Hepatic: Bilirubin less than 2 mg/dL Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 50 mL/min BUN no greater than 30 mg/dL Cardiovascular: No NYHA class III/IV status No active angina No myocardial infarction within 6 months No significant ventricular arrhythmia requiring medication No clinically significant conduction system abnormality Other: No serious intercurrent infection No nonmalignant medical illness that is uncontrolled or precludes study participation No psychiatric disorder that precludes informed consent No clinically significant auditory impairment No second malignancy within 5 years except: Basal cell skin cancer Carcinoma in situ of the cervix No pregnant or nursing women Negative pregnancy test required of fertile women Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: No prior chemotherapy or radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 1996-05; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Paul Kelsen, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States